CLINICAL TRIAL: NCT00335244
Title: A Phase III Single-Blind, Randomized, Placebo Controlled, Clinical Trial to Determine the Safety and Efficacy of Intravenous L-Citrulline Versus Placebo in Children Undergoing Cardiopulmonary Bypass
Brief Title: Intravenous L-Citrulline to Treat Children Undergoing Heart Bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 409; R01HL073317-01 (NIH); IRB# 060197
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Heart Defects, Congenital; Hypertension, Pulmonary
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intravenous L-citrulline
  Interventions: Drug: L-citrulline
- 2 (Placebo Comparator): Placebo of intravenous L-citrulline
  Interventions: Drug: Placebo of intravenous L-citrulline

INTERVENTIONS:
Drug: L-citrulline — 150mg bolus X 1 after initiation of cardiopulmonary bypass followed by continuous infusion of 9mg/kg/hr IV, starting 4 hours post bolus administration and ending at 48 hours continuous infusion or discharge from the PCCU
  Arms: 1
Drug: Placebo of intravenous L-citrulline — Placebo of intravenous L-citrulline
  Arms: 2

SUMMARY:
This clinical trial will determine the safety and effectiveness of intravenous L-citrulline in children undergoing cardiopulmonary bypass during heart surgery. Participants will be randomly assigned to either L-citrulline or a placebo (a substance that has no medicine in it).

Citrulline is a protein building block in the body that can convert into another substance, nitric oxide (NO), which controls blood pressure in the lungs. Increased blood pressure in the lungs can be an important surgical problem; it may also lead to problems following surgery, such as severe high blood pressure in the lungs (pulmonary hypertension), increased time spent on a breathing machine, and a longer stay in the intensive care unit (ICU). The hypothesis of this study is that perioperative supplementation with intravenous citrulline will increase plasma citrulline, arginine and NO metabolites and prevent elevations in the postoperative PVT leading to a decrease in the duration of postoperative invasive mechanical ventilation.

DETAILED DESCRIPTION:
Increased pulmonary vascular tone (PVT) can complicate the postoperative course of the following five surgical procedures for congenital heart defects: 1) unrestrictive ventricular septal defect (VSD) repair; 2) atrioventricular septal (AVSD) repair; 3) arterial switch procedure for transposition of the great arteries (TGA); 4) bidirectional Glenn shunt procedure; and 5) Fontan procedure for single ventricle lesions. PVT is partially controlled by NO. Arginine, the precursor to NO, is a product of the urea cycle. Preliminary data have been presented regarding 169 infants and children who have undergone one of six previous surgical procedures. It was found that urea cycle function and plasma arginine levels were significantly decreased in all participants. Furthermore, participants with increased PVT had significantly lower arginine levels compared to participants with normal PVT. Finally, a genetic single nucleotide polymorphism (SNP) in the rate limiting urea cycle enzyme (carbamyl phosphate synthetase I [CPSl T1405N]) appeared to affect postoperative plasma arginine levels and PVT. The hypothesis is that genetic polymorphisms in the rate limiting urea cycle enzyme CPSl, and other important enzymes in the urea cycle, influence the availability of NO precursors. It is further hypothesized that perioperative enhancement of urea cycle function with the key urea cycle intermediate (citrulline) will increase plasma arginine and NO metabolites and prevent elevations in PVT.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiopulmonary bypass surgery with 1 of the following 5 procedures:

  1. AVSD repair
  2. VSD repair
  3. Bidirectional Glenn
  4. Modified Fontan
  5. Arterial switch

Exclusion Criteria:

* Pulmonary artery or vein abnormalities not being addressed surgically
* Preoperative requirement for mechanical ventilation or intravenous inotrope support
* Any condition that might interfere with study objectives, as determined by the investigator
* Pregnant

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative mechanical ventilation in hours compared between treatment groups. | Measured in hours from the end of surgery until extubation

SECONDARY OUTCOMES:
Incidence of increased PVT (defined as a sustained mean pulmonary artery pressure greater than 20 mm Hg for at least 2 hours, measured during the first 48 hours | Measured in hours from the end of surgery until extubation
Postoperative intravenous inotrope score | Measured at 48 hours
Length and volume of chest tube drainage | Measured in hours from the end of surgery until removal of chest tubes
Length of ICU stay | Measured in hours from the end of surgery to discharge from ICU
Length of hospitalization | Measured from the day of surgery until discharge from hospital
Survival | Measured at 30 days post surgical repair

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick E. Barr, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States